CLINICAL TRIAL: NCT03548285
Title: A Phase II Study of Glottic Larynx Stereotactic Ablative Radiotherapy (LT-SABR) for Early-Stage Glottic Larynx Cancer
Brief Title: Stereotactic Ablative Radiotherapy for Early-stage Glottic Larynx Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, David Sher, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 122017-043
Record Dates: First submitted 2018-05-03; First posted 2018-06-07 (Actual); Results first posted 2025-04-25 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Glottic Carcinoma
MeSH Terms: interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SBRT Treatment (Experimental): Patients are all treated with stereotactic body radiation therapy (SBRT), using either CyberKnife or volumetric modulated arc therapy (VMAT). Dosing is based on the patients' assessed risk. The two cohorts are low risk and moderate risk.
  Low-risk is defined by:
  * Planning target volume (PTV) less than 10 cc, AND
  * No reported smoking within 1 month from registration
  Radiation Therapy will be delivered twice per week for 5 fractions (total 42.5 Gy)- this provides both an adequate tumoricidal dose, and a limited dose to normal tissue.
  Moderate-risk is defined by:
  * Planning target volume (PTV) greater than or equal to 10 cc, OR
  * Smoking within 1 month from registration (no more than 1 pack per day)
  Radiation Therapy will be delivered daily for 16 fraction (total 58.08 Gy)
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Stereotactic ablative radiotherapy (SABR), also known as stereotactic body radiation therapy (SBRT)

SUMMARY:
This is a prospective study to determine the local control and quality-of-life outcomes of using SBRT for early-stage glottic larynx cancer.

DETAILED DESCRIPTION:
SBRT treatment will be delivered to patients diagnosed with stage I-II glottic larynx cancer twice per week for 5 fractions (42.5 Gy cohort, low-risk) or daily for 16 fractions (58.08 Gy cohort, moderate-risk).

Low-risk is defined by:

* Planning target volume (PTV) less than 10 cc, AND
* No reported smoking within 1 month from registration

Moderate-risk is defined by:

* Planning target volume (PTV) greater than or equal to 10 cc, OR
* Smoking within 1 month from registration (no more than 1 pack per day)

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically-proven diagnosis of squamous cell carcinoma in situ, squamous cell carcinoma or squamous cell variants (sarcomatoid, verrucous, basaloid, and papillary subtypes) involving the glottic larynx.
2. Clinical stage I-II (American Joint Committee on Cancer AJCC, 7th edition) with direct laryngoscopy showing no evidence of greater than stage II true glottic larynx cancer and PET/CT or CT neck showing no evidence of regional disease.
3. Age ≥ 18 years.
4. ECOG Performance Status 0-2
5. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   5.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
6. Negative serum or urine pregnancy test within 2 weeks before registration for women of childbearing potential.
7. Ability to understand and the willingness to sign a written informed consent.
8. Patients with cognitive impairment or other limited decision making capacity with the ability to understand and willingly sign written informed consent or have the consent signed by a designated legally authorized representative (LAR)

Exclusion Criteria:

1. AJCC stage III or stage IV larynx cancer
2. Involvement of the arytenoid cartilage beyond the vocal process.
3. Prior chemotherapy for treatment of the targeted larynx lesion
4. Synchronous primaries in the head and neck
5. Prior radiotherapy to the region of the study cancer that would result in overlap of radiation fields.
6. Subjects smoking in excess of 1 pack of cigarettes per day.
7. Subjects may not be receiving any other investigational agents.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2024-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Sher, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Zhao B, Park YK, Gu X, Reynolds R, Timmerman R, Sher DJ. Surface guided motion management in glottic larynx stereotactic body radiation therapy. Radiother Oncol. 2020 Dec;153:236-242. doi: 10.1016/j.radonc.2020.08.027. Epub 2020 Sep 3. PMID 32890609

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Receiving SBRT Treatment: Radiation therapy: Stereotactic ablative radiotherapy (SABR), also known as stereotactic body radiation therapy (SBRT) Early-stage larynx cancer patients; all patients received SBRT (study treatment) at one of two different dose levels based on cohort (determined by whether the patient was low or moderate risk). The treatment fields are identical in both cohorts, and are expected to have the same patterns-of-failure. The dosing of these patients is not experimental and therefore was not a factor in analysis: all patients were analyzed together, as all received the same experimental treatment (SBRT). The biologically effective dose of this regimen is identical according to EQD2 (equivalent dose in 2 Gray fractions) analysis; in 5 fractions, the dose was equivalent to 65.52 Gy, and in 16 fractions, the dose was equivalent to 65.28 Gy. Therefore the biological impact of both regimens was the same, and this equivalence is why we analyzed the AE's together. The only potential difference between these dosing regimens is in late effects (1 year and after), but we saw no grade 2 or higher adverse events in either cohort, eliminating the need to report out late adverse events separately.
Period: Overall Study
Arm/Group | Patients Receiving SBRT Treatment
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Early stage larynx cancer patients receiving SBRT; additional details in participant flow
Groups:
- Patients Receiving SBRT: All patients on the clinical trial are receiving SBRT. Early-stage larynx cancer patients; all patients received SBRT (study treatment) at one of two different dose levels based on cohort (determined by whether the patient was low or moderate risk). The treatment fields are identical in both cohorts, and are expected to have the same patterns-of-failure. The dosing of these patients is not experimental and therefore was not a factor in analysis: all patients were analyzed together, as all received the same experimental treatment (SBRT). The biologically effective dose of this regimen is identical according to EQD2 (equivalent dose in 2 Gray fractions) analysis; in 5 fractions, the dose was equivalent to 65.52 Gy, and in 16 fractions, the dose was equivalent to 65.28 Gy. Therefore the biological impact of both regimens was the same, and this equivalence is why we analyzed the AE's together. The only potential difference between these dosing regimens is in late effects (1 year and after), but we saw no grade 2 or higher adverse events in either cohort, eliminating the need to report out late adverse events separately.
Arm/Group | Patients Receiving SBRT
Number analyzed (Participants) | 25
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Age of patients | 72 [65 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 19
  More than one race | 0
  Unknown or Not Reported | 2
Smoking [Number; unit: participants]
  None | 8
  Previous | 16
  Active | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Local Failure Following SABR Treatment of Early Glottic Larynx Cancers
Description: Local failure is defined as biopsy-proven tumor anywhere on the true vocal cords.
Time Frame: 2 years
Measure: Number; unit: participants
Groups:
- All Patients: All patients on the clinical trial.
Arm/Group | All Patients
Number analyzed (Participants) | 25
participants | 2

2. Secondary Outcome: Voice-quality Score Following Treatment With SABR
Description: Voice Handicap Index (VHI) voice-quality score to monitor changes in self-perception of voice handicap before and after treatment.
  0-30 Mild Minimal amount of handicap 31-60 Moderate handicap 60-120 Severe handicap
Time Frame: From baseline to 2 years post-treatment
Population: Participants who were able and willing to fill out PROs
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- 1M Follow up: One month follow up timepoint
- 6M Follow up: Six month follow up timepoint
- 12M Follow up: Twelve month follow up timepoint
- 24M Follow Up: Twenty-four month follow up timepoint
- Baseline: Baseline Timepoint
Arm/Group | 1M Follow up | 6M Follow up | 12M Follow up | 24M Follow Up | Baseline
Number analyzed (Participants) | 22 | 18 | 18 | 11 | 21
score on a scale | 28.5 [8 to 48] | 4 [0 to 12] | 7.5 [0 to 12] | 7.5 [0 to 12] | 57 [32 to 69]

3. Secondary Outcome: Number of Patients With Grade 3-5 Acute and Late Toxicities Following Treatment With SABR
Description: Number of patients with grade 3-5 acute (start of treatment through 90 days from the completion of treatment) and late (after 90 days from the completion of treatment) adverse events, according to NCI's Common Terminology Criteria for Adverse Events (CTCAE) v4.0 toxicity criteria.
Time Frame: 90 days, 3 years
Measure: Number; unit: participants
Arm/Group | All Patients
Number analyzed (Participants) | 25
participants
  Acute | 6
  Late | 19

4. Secondary Outcome: Health-related Quality of Life Following Treatment With SABR.
Description: Average patient visual analogue scale score (derived from EQ-5D) at baseline, 6, 12, and 24 months from the end of treatment
  The Visual Analogue Score (VAS) of the EQ-5D is a visual scale from 0-100, with 100 being perfect health, where patients can mark their perceived health. Researchers can then take the average score across all patients for each timepoint.
Time Frame: From baseline to 2 years post-treatment
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Patients Receiving SBRT Treatment
Number analyzed (Participants) | 25
score on a scale
  Baseline | 78 [0 to 100]
  6 Months | 86.2 [0 to 100]
  12 Months | 83.2 [0 to 100]
  24 Months | 85.5 [0 to 100]

5. Secondary Outcome: Percentage of Participants With Locoregional Failure Following SABR With Death as a Competing Risk
Description: Specifically, the 2-year cumulative risk of biopsy-proven recurrence anywhere in the larynx or neck following SABR. Recurrence in this context includes biopsy-proven cancer anywhere in the supraglottic, glottic, or subglottic larynx, as well as any malignant lymph node in the cervical or supraclavicular lymph nodes.
Time Frame: 2 years
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 25
Percentage of participants
  2 Years | 8 [3 to 24]
  1 Year | 4 [0.8 to 20]

6. Secondary Outcome: Overall Survival
Description: Overall survival
Time Frame: 2 years
Measure: Number; unit: patients
Arm/Group | All Patients
Number analyzed (Participants) | 25
patients
  Passed | 4
  Survival | 21

7. Secondary Outcome: Percentage of Patient Population With Regional Failure and Distant Metastasis
Description: With death and prior locoregional failure as competing risks
Time Frame: 2 years
Measure: Number; unit: Percentage of participants
Arm/Group | All Patients
Number analyzed (Participants) | 25
Percentage of participants
  2-year regional recurrence | 8
  2-year distant metastasis | 8

8. Secondary Outcome: Laryngectomy-free Survival
Description: Laryngectomy-free survival probability at 2 years
Time Frame: 2 years
Measure: Number; unit: Percentage of patients with LFS at 2 yrs
Arm/Group | All Patients
Number analyzed (Participants) | 25
Percentage of patients with LFS at 2 yrs | 88

ADVERSE EVENTS:
Time Frame: From baseline to 36M post treatment
Description: Adverse events were not collected separately based on dose. The AEs were evaluated with all patients together as one group.
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 4/25
Serious Adverse Events (participants affected / at risk) | 2/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=25)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (2)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2)
INR Increased (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=25)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (5)
Blurred vision (Eye disorders) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (4)
constipation (Gastrointestinal disorders) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 8 (9)
Creatinine increased (Investigations) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Dermatitis radiation (Injury, poisoning and procedural complications) | 2 (2)
diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 9 (13)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dysesthesia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 8 (8)
Dysphagia (Gastrointestinal disorders) | 6 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Edema (General disorders) | 1 (1)
Edema limb (General disorders) | 4 (4)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 9 (9)
Fever (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Odynophagia (Gastrointestinal disorders) | 5 (5)
Mucus Production (Gastrointestinal disorders) | 1 (1)
Voice fatigue (General disorders) | 1 (1)
Black stool (Gastrointestinal disorders) | 1 (1)
Headaches (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (2)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 12 (17)
hypercalcemia (Metabolism and nutrition disorders) | 1 (2)
Hypertension (Vascular disorders) | 17 (57)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypotension (Vascular disorders) | 1 (1)
Ear infection (Infections and infestations) | 1 (1)
Covid-19 (Infections and infestations) | 4 (4)
oral thrush (Infections and infestations) | 2 (2)
Cartilage tear (L ankle) (Injury, poisoning and procedural complications) | 1 (1)
Suprapubic catheter dysfunction (Injury, poisoning and procedural complications) | 1 (1)
torn meniscus L knee (Injury, poisoning and procedural complications) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Laryngeal edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Malignant neoplasm of prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
type II diabetes (Metabolism and nutrition disorders) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4)
hip pain (Musculoskeletal and connective tissue disorders) | 2 (2)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
nausea (Gastrointestinal disorders) | 2 (2)
Neck edema (General disorders) | 1 (1)
neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
polyp (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (3)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 (5)
urethral stricture (Renal and urinary disorders) | 1 (1)
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Salivary duct inflammation (Gastrointestinal disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (2)
erythema in left arytenoid (Skin and subcutaneous tissue disorders) | 1 (1)
Scalp lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 11 (15)
bladder prostate surgery (Surgical and medical procedures) | 1 (1)
Thick secretions (Gastrointestinal disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vocal cord inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-02-07): https://cdn.clinicaltrials.gov/large-docs/85/NCT03548285/Prot_SAP_000.pdf